CLINICAL TRIAL: NCT04616573
Title: A Prospective, Multi-center, Randomized, Masked, Controlled, Post-market Study Of Use Of The OMNI® Surgical System In Combination With Cataract Extraction In Open Angle Glaucoma (VERITA)
Brief Title: A Post-market Study Of Use Of The OMNI® Surgical System In Open Angle Glaucoma
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Sight Sciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 07024
Record Dates: First submitted 2020-10-30; First posted 2020-11-05 (Actual); Results first posted 2022-12-01 (Actual); Last update posted 2022-12-01 (Actual); Status verified 2022-11

CONDITIONS: Glaucoma, Open-Angle
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Ab-interno transluminal viscoelastic delivery with trabeculotomy using OMNI surgical System (Active Comparator): Ab-interno transluminal viscoelastic delivery with trabeculotomy using OMNI surgical System
  Interventions: Device: OMNI® Surgical System
- Ab-interno transluminal viscoelastic delivery using OMNI surgical System (Active Comparator): Ab-interno transluminal viscoelastic delivery using OMNI surgical System
  Interventions: Device: OMNI® Surgical System
- iStent Inject implantation (Active Comparator): iStent Inject implantation using the iStent device
  Interventions: Device: iStent inject

INTERVENTIONS:
Device: OMNI® Surgical System — Ab-interno transluminal viscoelastic delivery and trabeculotomy performed with the OMNI Surgical System
  Arms: Ab-interno transluminal viscoelastic delivery using OMNI surgical System; Ab-interno transluminal viscoelastic delivery with trabeculotomy using OMNI surgical System
Device: iStent inject — Trabecular meshwork implantation
  Arms: iStent Inject implantation

SUMMARY:
To prospectively compare the clinical effect of the OMNI surgical system in eyes with Open Angle Glaucoma.

DETAILED DESCRIPTION:
First, to prospectively compare the clinical effect of the transluminal viscoelastic delivery and trabeculotomy using the OMNI Surgical System to the iStent Inject used with Cataract Extraction in eyes with open angle glaucoma (OAG) and second, to prospectively compare the clinical effect of the transluminal viscoelastic delivery using the OMNI Surgical System to the iStent Inject used with Cataract Extraction in eyes with open angle glaucoma (OAG)

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, 22 years or older
* Visually significant cataract
* Mild to moderate open angle glaucoma
* On 1-5 IOP-lowering medications
* Potential of good best corrected visual acuity post cataract extraction, in the investigator's judgment
* Able and willing to comply with the protocol, including all follow-up visits.
* Understand and sign the informed consent.

Exclusion Criteria:

* Any of the following prior treatments for glaucoma:

  * Laser trabeculoplasty ≤3 months prior to baseline
  * Implanted with iStent (All types), Cypass, Xen, Express, glaucoma draining device/valve, or Hydrus Device
  * Prior canaloplasty, goniotomy, trabeculotomy, trabeculectomy, ECP or CPC
* Acute angle closure, normal tension, traumatic, congenital, malignant, uveitic, neovascular or severe glaucoma as documented in subjects' medical record.
* Concurrent ocular pathology or systemic medical condition which, in the Investigator's judgment, would either place the subject at increased risk of complications, contraindicate surgery, place the subject at risk of significant vision loss during the study period (e.g., wet AMD, corneal edema, Fuch's dystrophy, active intraocular infection or inflammation within 30 days prior to Screening Visit, etc.), or interfere with compliance to elements of the study protocol (e.g., returning to Investigator's office for follow-up visits).
* Participation (≤ 30 days prior to baseline) in an interventional trial which could have a potential effect on the study outcome, as determined by the study investigator
* Women of childbearing potential if they are currently pregnant or intend to become pregnant during the study period; are breast-feeding; or are not in agreement to use adequate birth control methods to prevent pregnancy throughout the study.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2020-11-13 (Actual); Primary Completion 2021-01-20 (Actual); Study Completion 2021-01-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kavita Dhamdhere, MD, PhD, Study Chair — Sight Sciences, Inc.
Locations (2):
- United States (2):
  - Eye Center South, Dothan, Alabama
  - Eye Associates and SurgiCenter of Vineland, Vineland, New Jersey

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ab-interno Transluminal Viscoelastic Delivery With Trabeculotomy Using OMNI Surgical System | Ab-interno Transluminal Viscoelastic Delivery Using OMNI Surgical System | iStent Inject Implantation
Started | 1 | 0 | 0
Completed | 0 | 0 | 0
Not Completed | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Only one subject was treated in the study. Study terminated early. No data to report for the other arms
Groups:
- Total: Total of all reporting groups
Arm/Group | Ab-interno Transluminal Viscoelastic Delivery With Trabeculotomy Using OMNI Surgical System | Ab-interno Transluminal Viscoelastic Delivery Using OMNI Surgical System | iStent Inject Implantation | Total
Number analyzed (Participants) | 1 | 0 | 0 | 1
Age, Continuous [Mean (Full Range); unit: years] | 66 |  |  | 66
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 1 |  |  | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 |  |  | 0
  Not Hispanic or Latino | 1 |  |  | 1
  Unknown or Not Reported | 0 |  |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  |  | 0
  Asian | 0 |  |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  |  | 0
  Black or African American | 0 |  |  | 0
  White | 1 |  |  | 1
  More than one race | 0 |  |  | 0
  Unknown or Not Reported | 0 |  |  | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Unmedicated Diurnal Intraocular Pressure (DIOP)
Description: The trial was terminated early after randomization and treatment of one subject who was exited from the study after 1 week of follow up. No meaningful conclusions or results were obtained due to early termination after the treatment of one subject.
Time Frame: 1 week
Population: No subjects were analyzed is for the 2 arms that did not have any subjects treated in the study.
Measure: Number; unit: mmHg
Arm/Group | Ab-interno Transluminal Viscoelastic Delivery With Trabeculotomy Using OMNI Surgical System | Ab-interno Transluminal Viscoelastic Delivery Using OMNI Surgical System | iStent Inject Implantation
Number analyzed (Participants) | 1 | 0 | 0
mmHg | 13.3 |  |

2. Secondary Outcome: Eyes With a ≥ 20% Decrease in Unmedicated Mean Diurnal Intraocular Pressure (DIOP) From Baseline
Description: as for outcome 1
Time Frame: 1 week
Population: The number analyzed is zero for the 2 arms of the study that did not treat any subjects/Eyes
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Ab-interno Transluminal Viscoelastic Delivery With Trabeculotomy Using OMNI Surgical System | Ab-interno Transluminal Viscoelastic Delivery Using OMNI Surgical System | iStent Inject Implantation
Number analyzed (Participants) | 1 | 0 | 0
Number analyzed (Eyes) | 1 | 0 | 0
Eyes | 1 |  |

3. Secondary Outcome: Eyes With Unmedicated Diurnal Intraocular Pressure (DIOP) Between 6 and 18 mmHg Inclusive
Description: as for outcome 1
Time Frame: 1 week
Population: The number analyzed is zero for 2 arms in the study which had no subjects treated
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Ab-interno Transluminal Viscoelastic Delivery With Trabeculotomy Using OMNI Surgical System | Ab-interno Transluminal Viscoelastic Delivery Using OMNI Surgical System | iStent Inject Implantation
Number analyzed (Participants) | 1 | 0 | 0
Number analyzed (Eyes) | 1 | 0 | 0
Eyes | 1 |  |

4. Secondary Outcome: Change in the Number of Ocular Hypotensive Medications Compared to Screening
Description: as for outcome 1
Time Frame: 1 week
Population: The number analyzed is zero for 2 arms in the study that did not have any treatments
Measure: Number; unit: number of hypotensive medications
Arm/Group | Ab-interno Transluminal Viscoelastic Delivery With Trabeculotomy Using OMNI Surgical System | Ab-interno Transluminal Viscoelastic Delivery Using OMNI Surgical System | iStent Inject Implantation
Number analyzed (Participants) | 1 | 0 | 0
number of hypotensive medications | 1 |  |

5. Secondary Outcome: Change in Unmedicated Diurnal Intraocular Pressure (DIOP) From Baseline
Description: as for outcome 1
Time Frame: 1 week
Population: The number analyzed is zero for 2 arms in the study that did not have any subjects treated.
Measure: Number; unit: mmHg
Arm/Group | Ab-interno Transluminal Viscoelastic Delivery With Trabeculotomy Using OMNI Surgical System | Ab-interno Transluminal Viscoelastic Delivery Using OMNI Surgical System | iStent Inject Implantation
Number analyzed (Participants) | 1 | 0 | 0
mmHg | 13.3 |  |

ADVERSE EVENTS:
Time Frame: 1 month
Description: There were no subjects enrolled in 2 arms that are showing zero "at risk" for AEs, SAEs or all cause mortality
Arm/Group | Ab-interno Transluminal Viscoelastic Delivery With Trabeculotomy Using OMNI Surgical System | Ab-interno Transluminal Viscoelastic Delivery Using OMNI Surgical System | iStent Inject Implantation
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 1/1 | 0/0 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ab-interno Transluminal Viscoelastic Delivery With Trabeculotomy Using OMNI Surgical System (N=1) | Ab-interno Transluminal Viscoelastic Delivery Using OMNI Surgical System (N=0) | iStent Inject Implantation (N=0)
Mild Blepharitis (Eye disorders) | 1 (1) | NA | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-31): https://cdn.clinicaltrials.gov/large-docs/73/NCT04616573/Prot_SAP_001.pdf